CLINICAL TRIAL: NCT00918151
Title: DiabCare Asia 2008 (Korea): A Cross-Sectional Survey to Evaluate Diabetes Management, Control, Complications, Psychosocial Aspects of Diabetic Patients in Asia & To Evaluate Perceptions and Practices of Physicians & Patients About Diabetes Management in Asia
Brief Title: A Survey to Evaluate Diabetes Management, Control, Chronic Complications, Psychosocial Aspects of Diabetic Subjects in Korea
Acronym: DiabCare Asia
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: INS-3781
Record Dates: First submitted 2009-06-09; First posted 2009-06-11 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Capillary or venous blood will be drawn for analysing HbA1c
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — Subject will only fill out a questionaire when entering the observational study

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate current status of diabetes management, control, and complications in diabetic subjects in Asia.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients registered in the particular centre for more than 12 months.
* Patients should have visited the centre at least once in the last 3-6 months apart from the initial visit.
* Patients willing to sign informed consent form.

Exclusion Criteria:

* Repetition of any patient as patients should not be included twice for any reason.
* Unwilling to participate or unable to comply with protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes mellitus (both type 1 and type 2) being treated at general hospitals, diabetes clinics and referral clinics will be selected according to the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1932 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Mean age of onset of type 1 and type 2 diabetes mellitus, respectively | at baseline visit/study start
Mean duration of treatment of type 2 diabetes mellitus. | at baseline visit/study start
Percentage of patients on insulin and Oral Anti-Diabetics Drugs (OADs) therapy, respectively | at baseline visit/study start
Mean duration of diabetes in type 1 and type 2 diabetic patients respectively | at baseline visit/study start
Mean FPG (fasting plasma glucose),PPG (post prandial glucose) and HbA1c of diabetic patients. | at baseline visit/study start
Percentage of diabetic patients with HbA1c target below 7.0% and below 6.5%, respectively | at baseline visit/study start
Percentage of diabetic patients having dyslipidemia and hypertension, cardiovascular complications, peripheral vascular disease, diabetic nephropathy and diabetic eye complications, respectively | at baseline visit/study start

SECONDARY OUTCOMES:
Patients' perception will be analysed through patient questionnaire measuring psychological well-being, quality of life and patients' compliant to treatment | at baseline visit/study start
Physician perception of diabetes and its management will be analysed through physician questionnaire measuring awareness about: HbA1c test and its goal, anti-diabetic treatment, barriers towards optimum diabetes control | at baseline visit/study start
Duration of diabetes associated with highest number of diabetic complications | at baseline visit/study start
Minimum duration of diabetes associated with 10% incidence of diabetic complications (CVD, nephropathy and retinopathy) | at baseline visit/study start

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Project Manager, Study Director — Novo Nordisk A/S
Locations (1):
- Seoul, South Korea

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com